CLINICAL TRIAL: NCT06449365
Title: Comparison of Intravenous V/S Nasal Atomizer Delivery of Midazolam for Conscious Sedation for No-scalpel Vasectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Tennessee Graduate School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: UTGSMIRB1123
Record Dates: First submitted 2024-02-28; First posted 2024-06-10 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Vasectomy; Sedation
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Intervention Model Description: randomized control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- midazolam delivery via intravenous (Active Comparator): normal sedation given via Intravenous route
  Interventions: Device: midazolam by nasal atomizer
- midazolam delivery via nasal atomizer (Active Comparator): normal sedation given via nasal atomizer
  Interventions: Drug: intravenous midazolam

INTERVENTIONS:
Device: midazolam by nasal atomizer — midazolam
  Other Names: midazolam
  Arms: midazolam delivery via intravenous
Drug: intravenous midazolam — midazolam
  Other Names: midazolam
  Arms: midazolam delivery via nasal atomizer

SUMMARY:
Purpose: This study compared administration of midazolam via intravenous route with nasal atomizer route for moderate sedation in an office-based vasectomy clinic.

DETAILED DESCRIPTION:
Purpose: This study compares administration of midazolam via intravenous route with nasal atomizer route for moderate sedation in an office-based vasectomy clinic.

Patients and methods: Patients will be randomly assigned to one of two groups: midazolam given via traditional intravenous route or midazolam via a nasal atomizer. Outcomes are patient perception of anxiety with the drug delivery method, discomfort with administration, pain during the procedure, and length of sedation effects. Medical personnel rated ease of use, efficacy, time to sedation and time to transport after procedure.

ELIGIBILITY:
Inclusion Criteria:

* all men who request no-scalpel vasectomy procedure

Exclusion Criteria:

* anyone not eligible for no-scalpel vasectomy procedure

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patient must be getting a non-scalpel vasectomy
Enrollment: 35 (Actual)
Dates: Start 2017-10-22 (Actual); Primary Completion 2020-08-07 (Actual); Study Completion 2020-08-07 (Actual)

PRIMARY OUTCOMES:
Patient Questionnaire (generated by institution) | 1 year
  comparison between groups

SECONDARY OUTCOMES:
Nursing Questionnaire (generated by institution) | 1 year
  comparison between groups

OTHER OUTCOMES:
Surgeon Questionnaire (generated by institution) | 1 year
  comparison between groups

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Ferris, Phd, Study Director — UTGSM
Locations (1):
- UTGSM, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
All data deidentified in a central database